CLINICAL TRIAL: NCT02499744
Title: Humidified High Flow Nasal Cannula Versus Nasal Intermittent Positive Ventilation in Neonates as Primary Respiratory Support:a Randomized Controlled Trial
Brief Title: Humidified High Flow Nasal Cannula Versus Nasal Intermittent Positive Ventilation in Neonates
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Gao WeiWei (Other)
Responsible Party: Sponsor-Investigator, Gao WeiWei, professor, Guangdong Women and Children Hospital
Organization: Guangdong Women and Children Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: GuangdongWCHHI
Record Dates: First submitted 2015-05-24; First posted 2015-07-16 (Estimated); Last update posted 2016-02-24 (Estimated); Status verified 2016-02

CONDITIONS: Respiratory Insufficiency
Keywords: NIPPV; HHFNC; RDS; neonate
MeSH Terms: conditions — Respiratory Insufficiency

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- HHFNC (Active Comparator): HHFNC is provided nasal cannula. Ventilator settings:fraction of inspired oxygen (FiO2):21-40%,flow:2-8(litre,L)/min,to maintain arterial blood hemoglobin oxygen saturation ( SaO2) at 90-95% The weaning process is left to the discretion of the attending physician.,when FiO2: 25%,flow:2(litre,L)/min.
  Interventions: Device: HHFNC
- NIPPV (Active Comparator): NIPPV is provided via binasal prongs. Ventilator settings:FiO2:21-40%,peak inspiratory pressure( PIP)：12-22cm H2O,positive and expiratory pressure(PEEP):5-7cm H2O,Rate:30-60 per minute to maintain SaO2 at 90-95%,The weaning process is left to the discretion of the attending physician,when FiO2: 25%,mean airway pressure (MAP):6cm H2O,R:30 per minute .
  Interventions: Device: NIPPV

INTERVENTIONS:
Device: NIPPV — For infants in the NIPPV-group who "fail"NIPPV (see definition below), need immediate intubation, a invasive "Rescue-Treatment" may be provided. The decision to attempt "Rescue-Treatment", the mode of respiratory support and the ventilator settings used are at the discretion of the attending clinician.
  Other Names: nasal intermittent postive pressure ventilaiton
  Arms: NIPPV
Device: HHFNC — For infants in the HHFNC-group who "fail"HHFNC (see definition below), need immediate intubation, a invasive "Rescue-Treatment" may be provided. The decision to attempt "Rescue-Treatment", the mode of respiratory support and the ventilator settings used are at the discretion of the attending clinician.
  Other Names: Humidified High Flow Nasal Cannula
  Arms: HHFNC

SUMMARY:
The investigators hypothesize that the Humidified High Flow Nasal Cannula(HHFNC) is effective and safe as primary respiratory support in neonate with respiratory distress syndrome(RDS). It is more convenient in HHFNC combined with kangaroo care.

DETAILED DESCRIPTION:
Today a new nursing principle proposed that is kangaroo care in neonate.Many study showed kangaroo care may reduce pain、decrease the respiratory and heart rate among preterm infant.The recently study show it benefit to Physical Growth and Neurodevelopment.

Respiratory failure remains a common problem in the neonatal intensive unit. As reported that early non-invasive ventilation is accompanied by significant improvement in subsequent lung development and alveolation.Nasal continuous positive airway pressure (NCPAP)、nasal intermittent positive pressure ventilation(NIPPV) and humidified high flow via nasal cannulas(HHFNC) are non-invasive ventilation models.But Unfortunately, NIPPV and NCPAP systems are not always easily applied or tolerated in the preterm infants.So it is not convenient in kangaroo care.Recently A meta analysis concluded that NIPPV is more effective than NCPAP in preterms respiratory diseases.Maybe the investigators can reason that NIPPV is effective than HHFNC,but there is limited data about the comparison of NIPPV and HHFNC as primary respiratory support in neonate.

The NIPPV group fail definition：1、FiO2>40%、MAP>10 centimeter water column (cm H2O),but SaO2<90%.2、significant abdominal distension.3、PaCO2>60 millimeter of mercury (mmHg)or partial pressure of arterial oxygen (PaO2)<45mmHg.4、severe apnea( definition:>6 episodes requiring stimulation in 6 hours or requiring >1 episodes of positive-pressure ventilation) 5.potential of hydrogen (PH)<7.2 The HHFNC group fail definition：1、FiO2>40%、flow>8 (litre,L)/min,but SaO2<90%.2、significant abdominal distension.3、PaCO2>60mmHg or PaO2<45mmHg.4、severe apnea 5.PH<7.2

ELIGIBILITY:
Inclusion Criteria:

1. Birth weight > 1000 grams and > 28 weeks gestation
2. have respiratory distress syndrome and need assistant ventilation

Exclusion Criteria:

1. Birth weight < 1000 grams
2. Estimated gestation < 28 weeks
3. infants have contraindications for use of non-invasive ventilation
4. Active air leak syndrome
5. Infants with abnormalities of the upper and lower airways; such as Pierre- Robin, Treacher-Collins, Goldenhar, choanal atresia or stenosis, cleft lip and/or palate, or
6. Infants with significant abdominal or respiratory malformations including trachea-esophageal fistula, intestinal atresia, omphalocele, gastroschisis, and congenital diaphragmatic hernia.

Max Age: 28 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 200 (Estimated)
Dates: Start 2016-02; Primary Completion 2017-05 (Estimated); Study Completion 2017-05 (Estimated)

PRIMARY OUTCOMES:
endotracheal intubation rate | 3 days
  endotracheal intubation rate assessed within 72 hours after extubation

SECONDARY OUTCOMES:
significant apnea | 7 days
  significant apnea measured by the Colin J definition:6 episodes requiring stimulation in 6 hours or requiring>1 episodes of positive -pressure ventilation
duration of non-invasive ventilation | 3 months
  the duration of ventilation measured by total non-invasive ventilation time in HHFNC and NIPPV groups
air leaks | 3 months
  air leak assessed by chest X-ray
full enteral feeding | 3 months
  full enteral feeding measured by total feeding dose above 120 ml per kilogram one day
Bronchopulmonary dysplasia | 3 months
  Bronchopulmonary dysplasia assessed by national institute of child health and human development(NICHD) definition
necrotizing enterocolitis | 3 months
  necrotizing enterocolitis assessed by abdominal X-ray and Bell classification
nasal trauma | 3 months
  nasal trauma measured by US national pressure Ulcer Advisory Panel(NPUAP)

OTHER OUTCOMES:
pain score | 3 months
  pain score assessed by neonatal infant pain scale (NIPS)
neurodevelopment | 3 months
  neurodevelopment assessed by Bayley scale

CONTACTS AND LOCATIONS:
Overall Officials: yang jie, doctor, Principal Investigator — Guangdong Women and Children Hospital

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- [Background] Chidambaram AG, Manjula S, Adhisivam B, Bhat BV. Effect of Kangaroo mother care in reducing pain due to heel prick among preterm neonates: a crossover trial. J Matern Fetal Neonatal Med. 2014 Mar;27(5):488-90. doi: 10.3109/14767058.2013.818974. Epub 2013 Jul 18. PMID 23796239
- [Background] Gathwala G, Singh B, Singh J. Effect of Kangaroo Mother Care on physical growth, breastfeeding and its acceptability. Trop Doct. 2010 Oct;40(4):199-202. doi: 10.1258/td.2010.090513. Epub 2010 Jul 28. PMID 20667921
- [Background] Padhi TR, Sareen D, Pradhan L, Jalali S, Sutar S, Das T, Modi RR, Behera UC. Evaluation of retinopathy of prematurity screening in reverse Kangaroo Mother Care: a pilot study. Eye (Lond). 2015 Apr;29(4):505-8. doi: 10.1038/eye.2014.340. Epub 2015 Jan 23. PMID 25613847
- [Background] Head LM. The effect of kangaroo care on neurodevelopmental outcomes in preterm infants. J Perinat Neonatal Nurs. 2014 Oct-Dec;28(4):290-9; quiz E3-4. doi: 10.1097/JPN.0000000000000062. PMID 25347107
- [Background] Thomson MA, Yoder BA, Winter VT, Martin H, Catland D, Siler-Khodr TM, Coalson JJ. Treatment of immature baboons for 28 days with early nasal continuous positive airway pressure. Am J Respir Crit Care Med. 2004 May 1;169(9):1054-62. doi: 10.1164/rccm.200309-1276OC. Epub 2004 Feb 12. PMID 14962819
- [Background] Shoemaker MT, Pierce MR, Yoder BA, DiGeronimo RJ. High flow nasal cannula versus nasal CPAP for neonatal respiratory disease: a retrospective study. J Perinatol. 2007 Feb;27(2):85-91. doi: 10.1038/sj.jp.7211647. PMID 17262040
- [Background] Davis PG, Lemyre B, de Paoli AG. Nasal intermittent positive pressure ventilation (NIPPV) versus nasal continuous positive airway pressure (NCPAP) for preterm neonates after extubation. Cochrane Database Syst Rev. 2001;(3):CD003212. doi: 10.1002/14651858.CD003212. PMID 11687052
- [Background] Woodhead DD, Lambert DK, Clark JM, Christensen RD. Comparing two methods of delivering high-flow gas therapy by nasal cannula following endotracheal extubation: a prospective, randomized, masked, crossover trial. J Perinatol. 2006 Aug;26(8):481-5. doi: 10.1038/sj.jp.7211543. Epub 2006 May 25. PMID 16724119